CLINICAL TRIAL: NCT06146127
Title: Precision Medicine for Combined Hepatocellular-Cholangiocarcinoma
Acronym: PREMED-CHC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Inserm U955 (Other)
Responsible Party: Principal Investigator, Julien Calderaro, Full Professor, Inserm U955
Other Study IDs: PREMED-CHC
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Liver Cancer
Keywords: liver; cancer; precision medicine
MeSH Terms: conditions — Liver Neoplasms; Neoplasms | interventions — Immunophenotyping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — frozen and ffpe samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Combined hepatocellular cholangiocarcinoma
  Interventions: Other: phenotyping
- hepatocellular carcinoma
  Interventions: Other: phenotyping
- cholangiocarcinoma
  Interventions: Other: phenotyping

INTERVENTIONS:
Other: phenotyping — Large scale molecular phenotyping

SUMMARY:
Our project is a large-scale characterisation of cHCC-CCA will allow us to determine which subsets harbor actionable gene alterations. We will also aim to improve diagnosis of this tumor type by the use of immunohistochemical biomarkers and the development of deep-learning based models able to help cHCC-CCA diagnosis. This will represent an important step towards precision medicine for the patients with this highly aggressive malignancy.

DETAILED DESCRIPTION:
* Scientific background Combined hepatocellular-cholangiocarcinoma (cHCC-CCA) is a rare liver cancer characterized by a dual hepatocytic and biliary differentiation. It is resistant to conventional anti-cancer treatments and there is currently no effective systemic therapy available. Inter-observer agreement for diagnosis of cHCC-CCA is low, even among expert pathologists, and the development of clinical trials remain thus challenging. The molecular mechanisms that drive its progression also remain under-investigated.
* Project objectives and brief description of the methods which will be used to achieve them We aim to perform an integrative molecular, immune and phenotypical study of cHCC-CCA that will allow the distinction of different tumor subgroups linked to particular actionable genetic/immune alterations. The development of immunohistochemical markers and artificial intelligence-based approaches is also likely to improve the diagnosis of cHCC-CCA.

A overall multicentric series of 357 cHCC-CCA samples, already available in our biobanks, will be investigated by means of gene and RNA sequencing, digital pathology and immunohistochemistry in order to build a morphomolecular classification of this tumor. Spatial transcriptomics and in situ proteomics will be performed to decipher the intra-tumor heterogeneity and identify biomarkers of the different subclasses. Finally, deep-learning based models will be developed in order to 1) improve the diagnosis of cHCC-CCA and 2) identify the morphological features linked to prognosis.

• Expected results This large-scale characterisation of cHCC-CCA will allow us to determine which subsets harbor actionable gene alterations. We will also aim to improve diagnosis of this tumor type by the use of immunohistochemical biomarkers and the development of deep-learning based models able to help cHCC-CCA diagnosis. This will represent an important step towards precision medicine for the patients with this highly aggressive malignancy.

ELIGIBILITY:
Inclusion Criteria:

histological diagnosis of combined tumor biological sample available

Exclusion Criteria:

unequivocal histological features

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adults
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2001-01-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosos | 3 yrs
  Tumor subgroups

CONTACTS AND LOCATIONS:
Overall Officials: Julien Calderaro, Principal Investigator — Inserm/APHP
Locations (1):
- Julien Calderaro, Créteil, France

IPD SHARING:
Plan to Share IPD: No